CLINICAL TRIAL: NCT06251713
Title: Feasibility of a Randomised Trial Comparing a Fluid-removal Guided by VeXUS Score With Usual Care in Patients With Acute Kidney Injury After Cardiac Surgery: a Pilot Randomised Trial.
Brief Title: Fluid-removal Guided by VeXUS Score With Usual Care in Patients With Acute Kidney Injury After Cardiac Surgery
Acronym: VeXUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL23_0891
Record Dates: First submitted 2024-01-15; First posted 2024-02-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury; Cardiac Surgery; Venous Congestion; Hemodynamic Stability
Keywords: Acute kidney injury; Cardiac surgery; Venous Congestion; VeXUS score; diuretic; fluid removal
MeSH Terms: conditions — Acute Kidney Injury; Hyperemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VeXUS score guided fluid management (Experimental): Fluid management:
  * Restrictive intake
  * Diuretic-induced fluid removal aiming for a diuresis of 2-4mL/Kg/h if VeXUS score > 1
  * During 24 to 48 hours
  Interventions: Other: VeXUS score guided fluid management strategy
- Usual care (Other): Fluid management:
  * Usual care
  * at the discretion of the attending physician
  Interventions: Other: Usual care

INTERVENTIONS:
Other: VeXUS score guided fluid management strategy — During the first 3 postoperative days, the VeXUS score is estimated daily by ultrasound. If VeXUS score >1, diuretic-induced fluid removal will be administred (target diuresis: 2-4mL/kg/h). The diuretic administration protocol is derived from the CARRESS HF study: bolus followed by a continuous administration of Furosemide with thiazide added based on preoperative diuretic administration status.
  To prevent hypokalaemia and dysnatremia, a protocol for potassium supplementation and intravenous administration of chloride serum or hypotonic perfusion is planned.
  Fluid removal will be suspended if severe metabolic disturbance (pH>7.55 with HCO3->40mmol/L or serum K+ <3 mmol/L or serum Na>150 mmol/L) or haemodynamic instability (hypoperfusion) with fluid responsiveness occurs. Regardless of the VeXUS score, diuretics will be introduced in case of pulmonary oedema.
  Haemodynamic status will be every 12 hours to detect side effects attributable to diuretic-induced fluid removal.
  Arms: VeXUS score guided fluid management
Other: Usual care — Fluid management will be at the discretion of attending physician, who will be blinded to the patient's VeXUS score status.
  Arms: Usual care

SUMMARY:
Acute kidney injury affects more than 30% of patients after cardiac surgery, and is associated with an excess in mortality. There is a clinical continuum between acute kidney injury (transient if <48h, persistent if >48h), the development of acute kidney and chronic renal failure. Each of these entities characterising renal recovery is associated with an increase in long-term morbidity and mortality. Fluid management in patients with acute kidney injury is challenging, as both hypovolaemia and hypervolaemia are detrimental. Venous congestion (reflecting intravascular hypervolaemia), is a well-established haemodynamic factor contributing to acute kidney injury after cardiac surgery. An ultrasound score, based on the venous doppler pattern explored in intra-abdominal organs, has recently been developed and is a better predictor of acute kidney injury than central venous pressure. Whether using the VeXUS score to guide fluid removal in haemodynamically stabilised patients could promote renal recovery after acute kidney injury remains to be investigated.

Before designing a large randomised trial to test such a strategy, its feasibility in a pilot randomised trial is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care unit admission within 72 hours of cardiac surgery with extracorporeal circulation
* Acute kidney injury defined by KDIGO criteria
* Vasoactive inotropic score <45 and capillary refill time <3s
* Informed written consent

Exclusion Criteria:

* Hypokalaemia <3.5mmol/L
* Hyponatremia<125mmol/L
* Hypernatremia >145mmol/L
* Metabolic alkalosis with pH >7.50
* Impossibility to measure capillary refill time
* Chronic liver disease
* Cirrhosis with portal hypertension
* Known thrombus of the inferior vena cava
* Mechanical circulatory assistance (ECMO or mono left ventricular assistance)
* Severe pre-operative chronic kidney disease (GFR < 30mL/min/1.73m2)
* Need for renal replacement therapy anticipated by the attending physician within 24 hours
* Known hypersensitivity to Furosemide and/or hydrochlorothiazide
* Severe allergy to wheat
* Patient already included in another interventional study with an exclusion period still in progress
* Pregnant, breast-feeding or women of childbearing age without suitable contraception
* Patients under guardianship, curatorship or safeguard of justice
* Patients under psychiatric care
* Patients not affiliated to a social security scheme or beneficiaries of a similar scheme

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Randomized controlled study feasibility | 48 hours after the inclusion
  Percentage of patients recruited without deviations from the protocol (number of patients included per month) at the end of the recruitment and follow-up period, i.e. the number of patients who received the full initial treatment (48 hours) in accordance with the interventional protocol out of the number of patients eligible for the study.

SECONDARY OUTCOMES:
Description of the "standard practice" group | 48 hours after the inclusion
  The standard practice groupe will be describe. The description will be based on the number of patients concerned by the administration of diuretics, molecule and dosage used, reason for the administration of diuretics, cumulative fluid balance.
Description of deviations from the protocol in the "intervention" group" | 48 hours after the inclusion
  To evaluation de faisability of the trial, the description of the deviations occurring in the intervention group will be based on the number of patients concerned, nature of the deviation from the protocol, cumulative fluid balance.
Venous congestion prevalence | Day 1
  Proportion of patients with VeXUS score >1 at the inclusion
Haemodynamic instability occurrence | Between inclusion and Hour 48 (H48)
  Occurrence of Mottling score>1 or capillary refill time>3s
Severe metabolic disturbance occurrence | Day 2
  Occurrence of serum potassium <3mmol/L, serum sodium >150 mmol/L, arterial pH>7.55 with HCO3->40mmol/L
Persistent acute Kidney Injury occurrence | 48 hours after the inclusion
  Description and comparison of the persistent acute Kidney Injury occurrence in the 2 groups
Use of Renal Replacement Therapy (RRT) occurrence | Day 30 (D30)
  Description and comparison of the RRT requirement in the 2 groups
Renal adverse events | Day 30 (D30)
  Description and comparison of the 2 groups for the composite criteria : death or Renal Replacement therapy dependence or creatinine > 200% baseline creatinine.
Acute kidney disease occurrence | Day 30 (D30)
  Description and comparison of the 2 groups for the composite criteria : albuminuria or GFR <60mL/min/1.73m or decrease of more than 35% in GFR.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Louis Pradel, Groupement Hospitalier Est, Hospices Civils de Lyon, Bron, Bron
  - Hopital cardiologique Louis Pradel, Bron

IPD SHARING:
Plan to Share IPD: No